CLINICAL TRIAL: NCT02041104
Title: Impact of Consumption of Beta-glucans on the Intestinal Microbiota and Glucose and Lipid Metabolism in a Population With Metabolic Syndrome
Brief Title: Impact of Consumption of Beta-glucans on the Intestinal Microbiota and Glucose and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mlinotest Zivilska Industrija d.d. (Industry)
Collaborators: University of Ljubljana (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLINOTEST/618-001
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome; Dyslipidemia; Obesity, Abdominal; Hyperglycemia; Hypertension
Keywords: Metabolic syndrome; 4 -week intervention; Randomised placebo controlled parallel study; Beta-glucans; Abdominal fat; Dyslipidemia; Insulin resistance; Hypertension; Gut Microbiota Composition; Oral Glucose Tolerance Test; Lipid Profile; Real-Time Polymerase Chain Reaction; Denaturating Gradient Gel Electrophoresis
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Obesity, Abdominal; Hyperglycemia; Hypertension; Insulin Resistance | interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bread with added beta-glucans (Experimental): Experimental food is bread with high amount of barley beta-glucans. Experimental bread contains approximately 3,4 % (w/w) beta-glucans. Participants will consume 6 g of beta-glucans daily (approximately 200 g of bread per day). Beta-glucans are natural polysaccharides found in grain endosperm and are mostly represented in oat and barley. Beta-glucans are linear homopolymers of D- glycopyranosyl residues with mixed linkage (1-4, 1-3)-β-D-glucans. Their molecular structure enable beta-glucans their functional action that mostly depends of their viscosity and solubility (1). Testing bread has integrated flour with high amount of barley beta-glucans (ReducholTM). Beta-glucans are concentrated in flour up to 15 % with dry milling, sieving and air classification of barley flour.
  Interventions: Dietary Supplement: Bread with added beta-glucans
- Bread without added beta-glucans (Placebo Comparator): Placebo bread without added barley beta-glucans in testing product.
  Interventions: Dietary Supplement: Placebo Comparator: Bread without added beta-glucans

INTERVENTIONS:
Dietary Supplement: Bread with added beta-glucans — Participants will daily consume bread with high content of beta-glucans. They will approximately consume 6 g beta-glucans per day in 200 g of bread. Intervention period will be 4 weeks. Meanwhile the participants will remain their usual eating habits except consuming any pro- or pre-biotics
  Arms: Bread with added beta-glucans
Dietary Supplement: Placebo Comparator: Bread without added beta-glucans — Participants will daily consume placebo bread without any added beta-glucans (approximately 200 g per day). Intervention period will be 4 weeks. Meanwhile the participants will remain their usual eating habits except consuming any pro- or pre-biotics.
  Arms: Bread without added beta-glucans

SUMMARY:
The purpose of this study is to investigate if daily consumption of barley beta-glucans effect lipid and glucose metabolism and alter intestinal microbiota composition in participants with metabolic syndrome or with high risk for metabolic syndrome development. It is assumed that 4-week intervention with beta-glucans will improve some clinical signs of metabolic syndrome and alter composition of intestinal microbiota. Variation in microbiota composition will be investigated with emphasis on Bacteroidetes and Firmicutes ratio. Furthermore it is presupposed that consumption of beta-glucans will stimulate growth of beneficial intestinal bacteria from genus Lactobacillus and Bifidobacteria and consequently effect production of short chain fatty acids in population with metabolic syndrome. Moreover it is presupposed that 4-week consumption of beta-glucans will have influence on glucose metabolism and will consequently improve insulin resistance within people with metabolic syndrome or high risk for metabolic syndrome development. It is assumed that 4-week consumption of beta-glucans will improve specific plasma lipid content in population with metabolic syndrome.

DETAILED DESCRIPTION:
In study it will be investigated whether daily consumption of barley beta-glucans integrated in bread product effects lipid and glucose metabolism and alter the composition of intestinal microbiota in a population with metabolic syndrome or with high risk for metabolic syndrome development. 70 participants with metabolic syndrome will be enrolled in study. Participants will daily consume 200 g of bread with high amount of beta-glucans.

Hypothesis:

1. 4- week consumption of beta-glucans alters composition of intestinal microbiota and changes ratio of bacteria from phylum Bacteroidetes and Firmicutes. Furthermore consumption of beta-glucans stimulates growth of beneficial intestinal bacteria from genus Lactobacillus and Bifidobacteria and consequently effects production of short chain fatty acids in population with metabolic syndrome.
2. 4- week consumption of beta-glucans has influence on glucose metabolism and consequently improves insulin resistance within people with metabolic syndrome.
3. 4 - week consumption of beta-glucans improves specific plasma lipid content in population with metabolic syndrome.

Study will be designed as double blind, randomised, placebo controlled clinical trial and performed regarding to CONSORT 2010 recommendations for randomised clinical trials. Patient enrollment will be performed in several community health centres in Slovenia in association with family medicine doctors. Appropriate patients with metabolic syndrome or with high risk for metabolic development will be suggested to participate in clinical trial. Candidates will be suggested to participate in a two month study. If there will not be recruited enough participants for two month study they will be suggested for participation in one month study. Candidates interested in participating in study will be informed about study design and terms and conditions of study by main investigator.

Study will be performed after successful recruitment of first 20 or more participants. Study will be performed three times, so that 70 participants will be recruited in complete study. Participants will consume bread with high beta-glucans content (around 3, 4 g beta-glucans per 100 g of bread) during 8 or 4 week period. Before beginning of study participants will have two week washout period without consuming any pre- and pro-biotics. They will remain their usual eating habits during study period except taking any antibiotics or pre- and pro-biotic. Participants will give blood and stool samples a day before intervention with barley beta-glucans. Blood sampling will involve oral glucose test for insulin resistance determination and sampling for specific lipid content determination. They will also have option to give a blood sample for genetic investigation of genes associated with lipid metabolism (apoE). Blood and stool sampling will be repeated day after intervention period. The same parameters as before intervention period except genetic analysis will be investigated. 72-hour dietary recall will be performed during intervention period individually to evaluate daily nutrient and energetic input of each participant.

ELIGIBILITY:
Inclusion Criteria are parameters used for metabolic syndrome determination according to International Diabetes Federation (IDF) consensus worldwide definition of Metabolic Syndrome:

Participant must have central obesity: defined as waist circumference ≥ 80 cm for European woman and ≥ 94 cm for European men. Beside central obesity candidates participating in this study must have total cholesterol concentration ≥ 5 mmol/l before entering the study.

Plus any two of the following four factors:

* HDL-cholesterol content: man ≤ 1,03 mmol/, women ≤ 1,23 mmol/l
* Triglycerides content ≥ 1,7 mmol/l
* Fasting blood glucose ≥ 5,6 mmol/l
* Hypertension: systolic blood pressure ≥ 130 mm Hg and diastolic blood pressure ≥ 85 mm Hg

If participant will have diagnosed metabolic syndrome and meet age criteria will be included in study.

Exclusion Criteria:

* Diabetes type II
* Thyroid disorder
* Kidney disorder
* Antibiotic treatment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Velikonja, PhD student, Principal Investigator — Mlinotest d.d. Zivilska Industrija; Rok Orel, M.D., D.Sc., Study Director — University Medical Centre Ljubljana; Gorazd Avgustin, UP, Study Director — University of Ljubljana
Locations (3):
- Slovenia (3):
  - Community Health Center Ajdovscina, Ajdovščina
  - Community Healt Center Ljubljana, Ljubljana
  - Community Health Center Franca Amrozica Postojna, Postojna

REFERENCES:
- [Background] (1) Izydorczyk MS,Dexter JE. Barley beta-glucans and arabinoxylans: Molecular structure, physicochemical properties, and uses in food products-a Review. Food Research International 41: 850-868, 2008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 81 participants were invited to trial trough national programme for metabolic disorder prevention and with help of family doctors. 30 participants were excluded due to personal reasons or because they did not meet inclusion criteria.
Groups:
- Bread With Added Beta-glucans: Experimental food was bread with a high amount of barley beta-glucans. Experimental bread contained approximately 3,4 g beta-glucans per 100 g of bread. Beta-glucans are natural polysaccharides found in grain endosperm and are mostly represented in oat and barley. Beta-glucans are linear homopolymers of D- glucopyranosyl residues with mixed linkage (1-4, 1-3)-β-D-glucans. Their molecular structure enables beta-glucans their functional action that mostly depends on their viscosity and solubility. For test bread preparation, we used flour with concentrated beta-glucans up to 15 %.
  Bread with added beta-glucans: Participants approximately consumed 6 g beta-glucans per day in 200 g of bread. The intervention period was 4 weeks long. Meanwhile, the participants remained their usual eating habits except consuming any pro- or pre-biotics
- Bread Without Added Beta-glucans: Placebo bread without added barley beta-glucans in the testing product.
  Placebo Comparator: Bread without added beta-glucans-Participants daily consumed placebo bread without any added beta-glucans (approximately 200 g bread per day). The intervention period was 4 weeks long. Meanwhile, the participants will remain their usual eating habits except consuming any pro- or pre-biotics.
Period: Overall Study
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Started | 28 | 23
Completed | 27 | 16
Not Completed | 1 | 7
Not completed — Lost to Follow-up | 1 | 4
Not completed — discomfort during OGTT | 0 | 3

BASELINE CHARACTERISTICS:
Population: The inclusion criteria for participants were as well diagnosed metabolic syndrome or high risk for metabolic syndrome development.
Groups:
- Bread With Added Beta-glucans: Experimental food was bread with a high amount of barley beta-glucans. Experimental bread contained approximately 3,4 g beta-glucans per 100 g of bread. Beta-glucans are natural polysaccharides found in grain endosperm and are mostly represented in oat and barley. Beta-glucans are linear homopolymers of D- glucopyranosyl residues with mixed linkage (1-4, 1-3)-β-D-glucans. Their molecular structure enables beta-glucans their functional action that mostly depends on their viscosity and solubility. Experimental bread was prepared with concentrated beta-glucans barley flour, containing up to 15 % of beta-glucans.
  Bread with added beta-glucans: Participants daily consumed bread with a high content of beta-glucans. They approximately consumed 6 g beta-glucans per day in 200 g of bread. The intervention period was 4 weeks long. Meanwhile, the participants remained their usual eating habits except consuming any pro- or pre-biotics
- Bread Without Added Beta-glucans: Placebo bread without added barley beta-glucans in the testing product.
  Placebo Comparator: Bread without added beta-glucans: Participants daily consumed placebo bread without any added beta-glucans (approximately 200 g bread per day). Intervention period will be 4 weeks. Meanwhile, the participants remained their usual eating habits except consuming any pro- or pre-biotics.
- Total: Total of all reporting groups
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans | Total
Number analyzed (Participants) | 27 | 16 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.93 (7.40) | 54.00 (8.07) | 52.07 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol Levels
Description: Before the intervention, total cholesterol levels were determined.
Time Frame: Baseline outcome measurement
Population: Total cholesterol levels were determined before diet intervention in both experimental groups.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 5.8 (1.01) | 5.9 (1.13)

2. Primary Outcome: HDL-cholesterol Levels
Description: HDL-cholesterol levels were determined before diet intervention.
Time Frame: Baseline measurement
Population: HDL-cholesterol levels were determined before diet intervention in both experimental groups.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 1.31 (0.44) | 1.51 (0.52)

3. Primary Outcome: LDL-cholesterol Levels
Description: LDL-cholesterol levels were determined before intervention
Time Frame: Baseline measurement
Population: LDL-cholesterol levels were determined in both experimental groups.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 3.99 (0.89) | 4.02 (0.91)

4. Primary Outcome: Determination of Composition of Intestinal Microbiota From Fecal Samples
Description: Fecal sampling for microbiologic analysis of microbiota composition: Composition of intestinal microbiota will be determined with a combination of two molecular techniques denaturating gradient gel electrophoresis (DGGE) and quantitative real time PCR (RT-PCR).
Time Frame: Outcome measurement at baseline
Population: We analyzed faecal samples of 40 participants from the test and control group. Since DGGE method is only qualitative measurement, the only measurements of RT-PCR are shown. Results are presented as relative numbers of specific bacteria group ((number of specific bacteria group / all bacteria)*100).
Measure: Mean (Standard Deviation); unit: % of bacteria
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 25 | 15
% of bacteria
  Bacteroides - Prevotella group | 7.95 (6.61) | 6.94 (3.57)
  Clostridium leptum group (cluster IV) | 28.22 (11.33) | 29.58 (11.90)
  Clostridium coccoides group (cluster XIVa) | 51.02 (22.91) | 58.03 (23.79)
  Enterobacteriaceae group | 1.75 (5.65) | 1.81 (5.46)
  Bifidobacterium genus | 0.62 (0.91) | 0.54 (1.15)
  Lactobacillus genus | 0.03 (0.06) | 0.31 (0.06)

5. Primary Outcome: Oral Glucose Tolerance Test (OGTT) for Insulin Resistance Determination (Outcome Measures of Plasma Insulin Concentrations)
Description: Pharmacokinetic outcome measures: Determination of insulin resistance with OGTT testing. Before and after oral consumption of 75 g of glucose, plasma insulin concentrations were measured at following times:
  0 min - before oral consumption of 75 g glucose 30 min, 60 min and 120 min - after oral consumption of 75 g glucose
Time Frame: OGTT measurements performed before dietary intervention
Population: In a population with metabolic syndrome or with high risk for metabolic syndrome development, OGTT was performed before dietary intervention.
Measure: Mean (Standard Deviation); unit: uM/mL
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
uM/mL
  Insulin concentration at time 0 min | 8.85 (5.87) | 8.40 (7.75)
  Insulin concentration at time 30 min | 50.01 (36.05) | 39.60 (20.25)
  Insulin concentration at time 60 min | 64.95 (50.55) | 63.52 (28.09)
  Insulin concentration at time 120 min: number analyzed (Participants) | 26 | 15
  Insulin concentration at time 120 min | 50.15 (39.92) | 35.87 (12.04)

6. Primary Outcome: Oral Glucose Tolerance Test (OGTT) for Insulin Resistance Determination (Outcome Measures of Plasma Glucose Concentrations)
Description: Pharmacokinetic outcome measures: Determination of insulin resistance with OGTT testing. Before and after oral consumption of 75 g of glucose, plasma glucose concentrations were measured at following times:
  0 min - before oral consumption of 75 g glucose 30 min, 60 min and 120 min - after oral consumption of 75 g glucose
Time Frame: Outcome OGTT measurements performed before dietary intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: uM/mL
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
uM/mL
  Glucose concentration at time 0 min | 5.12 (0.85) | 5.00 (0.64)
  Glucose concentration at time 30 min | 7.67 (1.91) | 8.19 (1.60)
  Glucose concentration at time 60 min | 7.16 (2.75) | 7.46 (1.75)
  Glucose concentration at time 120 min: number analyzed (Participants) | 26 | 16
  Glucose concentration at time 120 min | 5.01 (1.12) | 4.92 (0.76)

7. Primary Outcome: Systolic and Diastolic Blood Pressure
Description: Before the intervention, systolic and diastolic blood pressure were measured. Measurement was performed to obtain parameters for metabolic syndrome definition. Measurements after dietary intervention weren't performed.
Time Frame: Outcome measurement at baseline.
Population: Systolic and diastolic blood pressure were measured before dietary intervention in a population with metabolic syndrome or with high risk for metabolic syndrome development.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mm Hg
  Systolic blood pressure | 135.56 (17.2) | 137.31 (12.26)
  Diastolic blood pressure | 82.11 (9.65) | 82.19 (5.73)

8. Primary Outcome: Determination of Concentration of Short Chain Fatty Acids (SCFA) Present in Fecal Samples
Description: Fecal sampling for SCFA determination: Content of specific SCFA (butyric acid, acetic acid and propionic acid) will be determined in fecal samples using Gas Chromatography.
Time Frame: Outcome measurement at baseline
Population: We analyzed the concentration of short fatty acids from faeces from 41 participants belonging to test (bread with added beta-glucans) or control group (bread without added beta-glucans).
Measure: Mean (Standard Deviation); unit: g/kg
Groups:
- Bread With Added Beta-glucans: Experimental food is bread with high amount of barley beta-glucans. Experimental bread contains approximately 3,4 % (w/w) beta-glucans. Participants will consume 6 g of beta-glucans daily (approximately 200 g of bread per day). Beta-glucans are natural polysaccharides found in grain endosperm and are mostly represented in oat and barley. Beta-glucans are linear homopolymers of D- glycopyranosyl residues with mixed linkage (1-4, 1-3)-β-D-glucans. Testing bread has integrated flour with high amount of barley beta-glucans (ReducholTM). Beta-glucans are concentrated in flour up to 15 % with dry milling, sieving and air classification of barley flour.
  Bread with added beta-glucans: Participants will daily consume bread with high content of beta-glucans. They will approximately consume 6 g beta-glucans per day in 200 g of bread. Intervention period will be 4 week.
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 25 | 16
g/kg
  Acetic acid concentration | 2.70 (1.58) | 3.58 (2.03)
  Propionic acid concentration | 0.91 (0.60) | 1.38 (0.9)
  Butyric acid concentration | 0.97 (0.71) | 1.48 (0.98)

9. Primary Outcome: Triglyceride Levels
Description: Before the diet intervention, triglyceride levels were measured in test (consuming bread with added beta glucans) and in control group (consuming bread without added beta glucans).
Time Frame: Outcome measure at baseline.
Population: Triglyceride levels were measured in participants with metabolic syndrome or with high risk for metabolic syndrome development.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 1.91 (1.23) | 1.62 (1.06)

10. Secondary Outcome: Determination of Composition of Intestinal Microbiota From Fecal Samples
Description: as for outcome 4
Time Frame: Outcome measurement after 4-week dietary intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % of bacteria
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 25 | 15
% of bacteria
  Bacteroides - Prevotella group | 10.88 (8.80) | 8.89 (5.70)
  Clostridium leptum group (cluster IV) | 26.41 (14.96) | 30.38 (11.78)
  Clostridium coccoides group (cluster XIVa) | 47.22 (21.95) | 52.99 (18.88)
  Enterobacteriaceae group | 0.79 (1.33) | 1.58 (3.59)
  Bifidobacterium genus | 1.07 (1.41) | 0.56 (0.58)
  Lactobacillus genus | 0.09 (0.36) | 0.10 (0.31)

11. Secondary Outcome: Determination of Concentration of Short Chain Fatty Acids (SCFA) Present in Fecal Samples
Description: as for outcome 8
Time Frame: Outcome measurement after 4-week dietary intervention
Population: We analyzed the concentration of short fatty acids from faeces from 41 participants belonging to test (bread with added beta-glucans) or control group (bread without added beta-glucans) after 4-week intervention period.
Measure: Mean (Standard Deviation); unit: g/kg
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 25 | 16
g/kg
  Acetic acid concentration | 2.93 (1.74) | 2.08 (1.03)
  Propionic acid concentration | 1.30 (0.90) | 1.52 (2.50)
  Butyric acid concentration | 1.12 (0.77) | 1.61 (2.09)

12. Secondary Outcome: LDL-cholesterol Levels
Description: LDL-cholesterol levels were determined after intervention
Time Frame: Outcome measurement after 4-week dietary intervention
Population: LDL-cholesterol levels were determined in both experimental groups.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 3.89 (0.89) | 4.02 (0.66)

13. Secondary Outcome: HDL-cholesterol Levels
Description: HDL-cholesterol levels were determined after diet intervention.
Time Frame: Outcome measurement after 4-week dietary intervention
Population: HDL-cholesterol levels were determined after diet intervention in participants with metabolic syndrome or with high risk for metabolic syndrome development.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 1.30 (0.43) | 1.47 (0.44)

14. Secondary Outcome: Triglyceride Levels
Description: After the diet intervention, triglyceride levels were measured in test (consuming bread with added beta glucans) and in control group (consuming bread without added beta glucans).
Time Frame: Outcome measure after 4-week dietary intervention.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 1.72 (1.04) | 1.50 (0.65)

15. Secondary Outcome: Total Cholesterol Levels
Description: After the intervention, total cholesterol levels were determined.
Time Frame: Outcome measurement after 4-week dietary intervention
Population: Total cholesterol levels were determined before diet intervention in both experimental groups.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
mmol/L | 5.54 (0.90) | 5.96 (0.85)

16. Secondary Outcome: Oral Glucose Tolerance Test (OGTT) for Insulin Resistance Determination (Outcome Measures of Plasma Glucose Concentrations)
Description: Pharmacokinetic outcome measures: Determination of insulin resistance with OGTT testing. Before and after oral consumption of 75 g of glucose, plasma glucose concentration measurements were performed at following times:
  0 min - before oral consumption of 75 g glucose 30 min, 60 min and 120 min - after oral consumption of 75 g glucose
Time Frame: Outcome OGTT measurements performed after 4-week dietary intervention
Population: In a population with metabolic syndrome or with high risk for metabolic syndrome development, OGTT was performed after dietary intervention.
Measure: Mean (Standard Deviation); unit: uM/mL
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
uM/mL
  Glucose concentration at time 0 min: number analyzed (Participants) | 26 | 16
  Glucose concentration at time 0 min | 4.98 (1.28) | 5.16 (0.71)
  Glucose concentration at time 30 min: number analyzed (Participants) | 23 | 13
  Glucose concentration at time 30 min | 6.81 (2.80) | 7.86 (3.14)
  Glucose concentration at time 60 min: number analyzed (Participants) | 23 | 12
  Glucose concentration at time 60 min | 6.81 (2.80) | 7.26 (3.39)
  Glucose concentration at time 120 min: number analyzed (Participants) | 23 | 12
  Glucose concentration at time 120 min | 5.29 (2.74) | 4.41 (1.98)

17. Secondary Outcome: Oral Glucose Tolerance Test (OGTT) for Insulin Resistance Determination (Outcome Measures of Plasma Insulin Concentrations)
Description: Pharmacokinetic outcome measures: Determination of insulin resistance with OGTT testing. Before and after oral consumption of 75 g of glucose, plasma insulin concentration measurements were performed at following times:
  0 min - before oral consumption of 75 g glucose 30 min, 60 min and 120 min - after oral consumption of 75 g glucose
Time Frame: Outcome OGTT measurements performed after 4-week dietary intervention
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: uM/mL
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
Number analyzed (Participants) | 27 | 16
uM/mL
  Insulin concentration at time 0 min: number analyzed (Participants) | 25 | 15
  Insulin concentration at time 0 min | 10.10 (5.64) | 9.27 (3.65)
  Insulin concentration at time 30 min: number analyzed (Participants) | 23 | 12
  Insulin concentration at time 30 min | 53.16 (29.05) | 47.07 (33.61)
  Insulin concentration at time 60 min: number analyzed (Participants) | 23 | 11
  Insulin concentration at time 60 min | 76.50 (60.54) | 67.85 (35.41)
  Insulin concentration at time 120 min: number analyzed (Participants) | 23 | 11
  Insulin concentration at time 120 min | 56.34 (48.07) | 43.5 (33.07)

ADVERSE EVENTS:
Time Frame: We performed a dietary intervention with high amounts of beta-glucans in test bread. We expected mild adverse events such as diarrhea or bloating, that disappear after stop consuming experimental bread. Regarding this, we collected adverse event data only during the interventional study (4 weeks).
Description: Adverse events were collected when participant detect some abnormalities during the intervention or during laboratory analysis.
  Participants could report adverse events any time by telephone to investigators performing clinical testing.
Arm/Group | Bread With Added Beta-glucans | Bread Without Added Beta-glucans
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/28 | 3/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bread With Added Beta-glucans (N=28) | Bread Without Added Beta-glucans (N=23)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — After few days of dietary trial, diarrhea appear to one participant in test group consuming bread with added beta-glucans.
Discomfort during OGTT analysis (Investigations) | 0 (0) | 3 (3) — Participants felt dizziness or sickness during first OGTT analysis. They refused to continue diet intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02041104/SAP_000.pdf
  • Study Protocol (2013-08-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT02041104/Prot_001.pdf